CLINICAL TRIAL: NCT03916562
Title: Toward a Mechanistic Understanding of Optimization Principles Underlying Hemiparetic Gait
Brief Title: Optimization Principles in Hemiparetic Gait
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James Finley, Assistant Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS-18-00533; R01HD091184 (NIH)
Record Dates: First submitted 2019-03-31; First posted 2019-04-16 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: Walking; Gait; Stability; Energetic cost
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: For this study, the investigators will recruit two separate groups of participants who will complete the study procedures in parallel. One group will be comprised of individuals post-stroke and the second group will be comprised of adults who have not had a stroke.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (Experimental): The investigators will determine how asymmetric walking constraints influence spatiotemporal coordination, energetic cost, and dynamic balance in healthy individuals. The investigators will manipulate spatiotemporal coordination using a special treadmill. Energetic cost will be quantified using expired gas analysis and inverse dynamic approaches. Stability will be evaluated by characterizing participants' ability to recover from unexpected perturbations.
  Interventions: Behavioral: Manipulation of spatiotemporal coordination during walking
- Post-stroke Participants (Experimental): The investigators will determine how different patterns of coordination during walking influence energetic cost and dynamic balance in people post-stroke. The investigators will manipulate coordination using a special treadmill. Energetic cost will be quantified using expired gas analysis and inverse dynamic approaches. Stability will be evaluated by characterizing participants' ability to recover from unexpected perturbations.
  Interventions: Behavioral: Manipulation of spatiotemporal coordination during walking

INTERVENTIONS:
Behavioral: Manipulation of spatiotemporal coordination during walking — A description of the intervention is included in the description of the study arms.

SUMMARY:
This project seeks to identify the how walking impairments in stroke survivors contribute to mobility deficits through the use of behavioral observations and computational models. The chosen approach integrates biomechanical analyses, physiological assessments and machine learning algorithms to explain how asymmetries during walking influence balance and the effort required to walk. Ultimately, the results of this work may lead to more personalized rehabilitation strategies to improve walking capacity and efficiency, and ultimately reduce fall risk in stroke survivors.

ELIGIBILITY:
Inclusion Criteria for Control Participants:

* No musculoskeletal injury or conditions that limit walking ability
* No history of neurological disorders or severe head trauma
* Absence of cognitive impairment as demonstrated by a Mini-Mental score greater than 24

Inclusion Criteria for Post-Stroke Participants

* Presence of unilateral brain lesion from a single stroke
* Weakness confined to one side
* Ability to walk on a treadmill for five minutes continuously without a cane or walker
* Absence of cognitive impairment as demonstrated by a Mini-Mental score greater than 24

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption (VO2) | At the beginning of study day one
  The investigators will use a metabolic cart to measure the rate of oxygen consumption (VO2) while participants walk at a fixed speed on a treadmill.
Correlation between oxygen consumption (VO2) and step length asymmetry | During study day one
  The investigators will use a metabolic cart to measure the rate of oxygen consumption (VO2) while participants walk at a fixed speed on a treadmill. VO2 will be measured in five trials where participants walk with different levels of step length asymmetry. This outcome will capture the relationship between measures of VO2 and step length asymmetry.
Angular momentum during walking | At the beginning of study day two
  Motion capture will be used to measure the kinematics of the body when participants respond to accelerations of the treadmill
Correlation between angular momentum and step length asymmetry during walking | During study day two
  Participants will complete five trials at different levels of step length asymmetry. During these trials, motion capture will be used to measure the kinematics of the body when participants respond to accelerations of the treadmill. This outcome measure will use data from all trials to determine the relationship between angular momentum and step length asymmetry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanchez N, Finley JM. Individual Differences in Locomotor Function Predict the Capacity to Reduce Asymmetry and Modify the Energetic Cost of Walking Poststroke. Neurorehabil Neural Repair. 2018 Aug;32(8):701-713. doi: 10.1177/1545968318787913. Epub 2018 Jul 12. PMID 29998788
- [Background] Liu C, Macedo L, Finley JM. Conservation of Reactive Stabilization Strategies in the Presence of Step Length Asymmetries During Walking. Front Hum Neurosci. 2018 Jun 27;12:251. doi: 10.3389/fnhum.2018.00251. eCollection 2018. PMID 29997488
- [Background] Sanchez N, Park S, Finley JM. Evidence of Energetic Optimization during Adaptation Differs for Metabolic, Mechanical, and Perceptual Estimates of Energetic Cost. Sci Rep. 2017 Aug 9;7(1):7682. doi: 10.1038/s41598-017-08147-y. PMID 28794494
- [Background] Finley JM, Bastian AJ. Associations Between Foot Placement Asymmetries and Metabolic Cost of Transport in Hemiparetic Gait. Neurorehabil Neural Repair. 2017 Feb;31(2):168-177. doi: 10.1177/1545968316675428. Epub 2016 Oct 22. PMID 27798378
- [Background] Finley JM, Long A, Bastian AJ, Torres-Oviedo G. Spatial and Temporal Control Contribute to Step Length Asymmetry During Split-Belt Adaptation and Hemiparetic Gait. Neurorehabil Neural Repair. 2015 Sep;29(8):786-95. doi: 10.1177/1545968314567149. Epub 2015 Jan 14. PMID 25589580
- [Derived] Park S, Liu C, Sanchez N, Tilson JK, Mulroy SJ, Finley JM. Using Biofeedback to Reduce Step Length Asymmetry Impairs Dynamic Balance in People Poststroke. Neurorehabil Neural Repair. 2021 Aug;35(8):738-749. doi: 10.1177/15459683211019346. Epub 2021 Jun 1. PMID 34060926